CLINICAL TRIAL: NCT04362592
Title: In-Utero Endoscopic Correction of Spina Bifida: Laparotomy-Assisted or Percutaneous
Brief Title: In-Utero Endoscopic Correction of Spina Bifida
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Southern California (Other)
Collaborators: USFetus (Other)
Responsible Party: Principal Investigator, Ramen Chmait, Assistant Professor, University of Southern California
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: HS-05-00374
Record Dates: First submitted 2020-03-24; First posted 2020-04-27 (Actual); Last update posted 2025-03-28 (Actual); Status verified 2025-03

CONDITIONS: Neural Tube Defects; Spina Bifida; Myelomeningocele
MeSH Terms: conditions — Neural Tube Defects; Spinal Dysraphism; Meningomyelocele

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (2):
- Percutaneous Technique (Experimental): The percutaneous technique uses endoscopic scopes through the maternal skin and uterus to perform the surgery. A variation of the percutaneous technique is the mini-laparotomy technique, which uses an endoscopic scope through an incision on the abdomen, smaller than a laparotomy ("mini-laparotomy"), and smaller endoscopic scopes through the maternal skin and uterus to perform the surgery.
  Interventions: Device: In Utero Endoscopic Correction of Myelomeningocele IDE - Percutaneous Technique
- Laparotomy/Uterine Exteriorization Technique (Experimental): The laparotomy/uterine exteriorization technique consists of performing a laparotomy (incision into the abdominal cavity), exteriorizing the uterus, and using endoscopic scopes through the uterus to perform the correction.
  Interventions: Device: In Utero Endoscopic Correction of Myelomeningocele IDE - Laparotomy/Uterine Exteriorization Technique

INTERVENTIONS:
Device: In Utero Endoscopic Correction of Myelomeningocele IDE - Percutaneous Technique — The percutaneous approach uses endoscopes through a closed maternal abdomen and closed uterus to perform the spina bifida correction.
  Arms: Percutaneous Technique
Device: In Utero Endoscopic Correction of Myelomeningocele IDE - Laparotomy/Uterine Exteriorization Technique — The laparotomy/uterine exteriorization technique uses endoscopes through an open abdomen and closed, exteriorized uterus to perform the spina bifida correction.
  Arms: Laparotomy/Uterine Exteriorization Technique

SUMMARY:
The purpose of this study is to evaluate the feasibility and effectiveness of performing fetoscopic surgical correction of fetal spina bifida. Two surgical approaches will be utilized: the percutaneous technique versus the laparotomy/uterine exteriorization technique.

ELIGIBILITY:
Inclusion Criteria:

1. Myelomeningocele (including myeloschisis) at level T1 through S1 with hindbrain herniation. Lesion level and hindbrain herniation will be confirmed by MRI and ultrasonography.
2. Maternal age ≥18 years.
3. Gestational age of 19 to 27 6/7 weeks' gestation as determined by clinical information and evaluation of first ultrasound.
4. Balanced karyotype and/or normal mircoarray with written confirmation of culture results. Results by fluorescence in situ hybridization (FISH) will be acceptable if the patient is at 24 weeks or more.
5. Positive evaluation of social work consult indicating the patient is capable of consenting to the procedure and has the appropriate social support system to participate in the study.
6. Positive evaluation from pediatric neurology consult.
7. Willing to return to our center, or to a multi-disciplinary spina bifida clinic closer to their home for the 6, 12, 24, 30, 48, and 60 months follow-up evaluations.

Exclusion Criteria:

1. Multiple gestation
2. Insulin-dependent pregestational diabetes
3. Presence of a fetal anomaly not related to Chiari II Malformation. A fetal echocardiogram will be conducted before surgery and if the finding is abnormal, the patient will be excluded.
4. Fetal kyphosis of 30 degrees or more, assessed by ultrasound or MRI.
5. Presence of uterine cervical cerclage or history of incompetent cervix.
6. Placenta previa or placental abruption.
7. Short cervix < 25 mm measured by cervical ultrasound.
8. Obesity as defined by body mass index (BMI) of 40 or greater.
9. History of previous spontaneous singleton delivery prior to 37 weeks.
10. Maternal-fetal Rh isoimmunization, Kell sensitization or a history of neonatal alloimmune thrombocytopenia.
11. Maternal HIV or Hepatitis-B status positive because of the increased risk of transmission to the fetus during maternal-fetal surgery. If the patient's HIV or Hepatitis B status is unknown, the patient must be tested and found to have negative results before she can be enrolled.
12. Known Hepatitis-C positivity. If the patient's Hepatitis C status is unknown, she does not need to be screened.
13. Uterine anomaly such as large (greater than 6 cm) fibroids, cervical fibroids or multiple fibroids or Mullerian duct abnormality.
14. Other maternal medical condition which is a contraindication to surgery or anesthesia.
15. Patient does not have a support person (e.g., husband, partner, parents).
16. Inability to comply with the travel and follow-up requirements of the study.
17. Patient does not meet psychosocial criteria as determined by the social worker evaluation.
18. Participation in another intervention study that influences maternal and fetal morbidity and mortality.
19. Maternal hypertension as determined by the investigator, which would increase the risk of preeclampsia or preterm delivery (including, but not limited to: uncontrolled hypertension, chronic hypertension with end organ damage and new onset hypertension in current pregnancy).
20. Bicornuate uterus or any other uterine malformation the PI decides is not safe for surgery.
21. Nickel allergy.
22. Maternal request to undergo open fetal surgery for the antenatal correction of OSB at our institution primarily or after failed fetoscopic approach.
23. Known maternal hypersensitivity to bovine collagen or chondroitin materials.

Ages: 18 Years to 52 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — Gravid female
Enrollment: 110 (Estimated)
Dates: Start 2018-11-02 (Actual); Primary Completion 2026-06 (Estimated); Study Completion 2031-10-31 (Estimated)

PRIMARY OUTCOMES:
Ability to perform the endoscopic procedure | At time of surgery
  Successful fetoscopic closure of the defect

SECONDARY OUTCOMES:
Chiari II malformation reversal | Prior to delivery
  Reversal of hindbrain herniation on ultrasound and MRI

CONTACTS AND LOCATIONS:
Overall Officials: Ruben Quintero, MD, Principal Investigator — US Fetus; Ramen Chmait, MD, Principal Investigator — University of Southern California
Locations (2):
- United States (2):
  - Hollywood Presbyterian Medical Center, Los Angeles, California
  - Wellington Regional Medical Center, Wellington, Florida